CLINICAL TRIAL: NCT03724578
Title: Grape Seeds Versus Standard Measures for Prevention of Caries Incidence in Young Egyptian Adults: A Randomized Controlled Trial
Brief Title: Grape Seeds Versus Standard Measures for Prevention of Caries Incidence
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Omar Nader, Principal investigator, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 15102018
Record Dates: First submitted 2018-10-28; First posted 2018-10-30 (Actual); Last update posted 2018-11-02 (Actual); Status verified 2018-10

CONDITIONS: Dental Caries
MeSH Terms: conditions — Dental Caries | interventions — Anti-Infective Agents

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- standard preventive measures (Sham Comparator): the participants will only follow standard preventive measure twice a day brushing with fluoride toothpaste and flossing once a day
  Interventions: Drug: standard preventive measures
- antimicrobial and fluoride mouth wash (Active Comparator): participants will use mouth wash contains both chlorhexidine and fluoride in addition to standard preventive measures
  Interventions: Drug: antimicrobial and fluoride mouth wash
- grape seeds extract mouth wash (Experimental): the intervention is grape seeds extract mouth wash
  Interventions: Drug: Grape Seed Extract mouth wash

INTERVENTIONS:
Drug: Grape Seed Extract mouth wash — participants will use grape seeds extract mouth wash in addition to standard preventive measures
  Arms: grape seeds extract mouth wash
Drug: standard preventive measures — twice daily brushing with fluoride tooth pate and daily flossing
  Arms: standard preventive measures
Drug: antimicrobial and fluoride mouth wash — using chlorhexidine and fluoride containing mouth wash
  Arms: antimicrobial and fluoride mouth wash

SUMMARY:
The objective is to conduct an randomized controlled clinical trial to evaluate the effectiveness of grape seeds extract mouth wash in comparison with standard caries preventive measures for the prevention of new carious lesions in high caries risk patients.

This study will be designed to test the alternative hypothesis that using grape seed extract mouth wash in addition to standard preventive measures will show significant difference over using standard preventive measures alone in preventing incidence of new carious lesions in high caries risk patients

DETAILED DESCRIPTION:
Research Question:

In high caries risk patients, will the incorporation of grape seeds extract after using standard oral hygiene measures be beneficial in reducing caries risk and preventing the incidence of new carious lesions?

Intervention:

The study will be announced at the Faculty of Oral and Dental Medicine, Future University campus to encourage interested students to participate in the study.

Interested participants will be screened at Conservative Department clinic for eligibility. Eligible participants will be assessed using caries risk assessment tool (American Dental Association caries risk assessment form).

Eligible participants will be randomly divided into three groups 1st group will follow only standard preventive measures (tooth brushing twice a day with fluoride tooth paste and inter-dental flossing once daily), 2nd group will use grape seeds extract mouth wash beside standard preventive measure, and 3rd group will use antimicrobial mouthwash with fluoride beside standard preventive measure General operative procedures Before starting the study the eligible participants will undergo scaling and prophylaxis polishing, then any carious cavity, or defective restoration will be treated and filled with resin composite restoration.

New set of manual brushes and dental floss will be given to the participants, after they are properly trained for the correct brushing and flossing technique. The participants will be asked to brush their teeth twice a day with fluoride tooth paste and to clean their teeth inter-dentally with dental floss once a day every day till the end of the study. All the participants will undergo scaling and prophylaxis polishing at every recall visit Preparation of the grape seeds extract mouthwash

* Procedure of preparing Grape Seed Extract:

Grape seeds will be collected from grapes which are available in the market. These seeds will be dried under sunlight for 2 days, and then these seeds will be grounded with cold pressure technique. Ground grape seeds (100 gm) will be extracted with ethanol/water ratio of 70:30, vol/vol, by maceration method under stirring at 45 degree centigrade for 2 hours, then The extract will be filtered(19).

For the intervention 1 group Beside the standard preventive measures that the participants will be trained to follow, each patient will be given a bottle of grape seeds extract mouthwash.

The participants will be instructed to rinse 15 milliliter of the mouthwash twice a day after breakfast and before bedtime and to retain it in their mouth for one minute before expectorating it, and not to consume any food or drink for 30 minutes after the use of mouthwash(12).

For intervention 2 group The participants will be instructed to rinse 15 milliliter of the mouth twice a day after breakfast and before bedtime and to retain it in their mouth for one minute before expectorating it, and not to consume any food or drink for 30 minutes after the use of mouthwash. Participants will repeat this protocol for five days every month until the end of the study.

For the control group Participants in this group will follow only the standard preventive measures which is brushing twice a day after breakfast and before bed time and daily flossing inter-dentally before bed time.

In all study groups if any patient during the period of the study develops any carious cavity, the affected tooth will be treated immediately and restored with resin composite restoration.

Outcomes:

Visual inspection to detect presence or absence of new caries lesions will be done according to World Health Organization guidelines. Caries detection will be carried out after careful drying of the tooth surface using three-way syringe to facilitate detection of initial enamel lesions (white spot lesions). Also pits and fissure carious lesions will be detected using visual and tactile method. (26).

Sample size:

The aim of this study is to assess Incidence of new caries in Grape seeds versus standard measures for prevention of caries. Based on a previous paper by Zhang 2006(27) the difference in caries development (reduction by antimicrobial mouth wash) between at least 2 groups is 40%. Using power 80% and 5% significance level the investigators will need to study 22 in each group. This number is to be increased to a sample size of 26 to compensate for losses during follow up. Sample size calculation was achieved using PS: Power and Sample Size Calculation software Version 3.1.2 (Vanderbilt University, Nashville, Tennessee, USA

Recruitment:

Patients will be recruited by (S.K and O.N) from the students of Faculty of Oral and Dental medicine, Future University as the research is targeting young Egyptian adults, only the eligible participants will be chosen until reaching the target sample size.

-Baseline data collection: For every patient medical and dental history and caries risk assessment profile will be obtained. Examination chart will be filled by (O.N)

Outcome data collection:

Visual caries inspection and community periodontal index probe(28) will be used by the assessor (S.K and E.A) after 3 months, 6 months, 9 months and 1 year to evaluate the presence or absence of new caries lesions.

Patient retention:

The patient's phone number will be recorded in their charts and before every visit the patient will receive a reminder call by (O.N). If the patient did not answer, another appointment will be scheduled within a week.

No harms are expected as the intervention product is natural product and Considered as (generally recognized as safe) by The FDA (Food and Drug Administration Informed consent The trial will be explained to the patients by the principle investigator. The researcher will discuss the interventions and possible harms with patients and obtain written consent (in Arabic) from the patients willing to participate in the trial. An appendix of the consent form is attached to the protocol

Post-trial care All patients will complete their treatment by the same operator at the clinic of the Conservative Department. The participants will be followed up even after the trial ends (6 months follow up period) to treat patient's complaints and prevent any possible complications

ELIGIBILITY:
Inclusion Criteria:

* patients with High caries risk
* 18-25 years
* Males or females
* Medically free patients
* Patients approving to participate in the study

Exclusion Criteria:

* • Patients were on antibiotic therapy or corticosteroid therapy for 30 days before the examination

  * Patients had history of professional cleaning in the last 15 days
  * Patients with exposed pulp
  * Evidence of parafunctional habits
  * Patients with developmental dental anomalies
  * Patients undergoing or will start orthodontic treatment
  * Patients with removable prosthesis
  * Periapical Abscess or Fistula

Ages: 18 Years to 25 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 80 (Estimated)
Dates: Start 2019-01-01 (Estimated); Primary Completion 2020-02-01 (Estimated); Study Completion 2020-03-01 (Estimated)

PRIMARY OUTCOMES:
caries incidence | 12 months
  visual inspection of new carious lesions

IPD SHARING:
Plan to Share IPD: No